CLINICAL TRIAL: NCT02579681
Title: Single Country Study Assessing Cognition in Relapsing Remitting Multiple Sclerosis Patients Treated With BG00012
Brief Title: Study Assessing Cognition in Relapsing Remitting Multiple Sclerosis (RRMS) Patients Treated With BG00012
Acronym: StarTec
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITA-BGT-12-10389; 2013-001422-25 (EudraCT Number); 109MS410 (Other: Biogen)
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Cognition; Tecfidera; RRMS; BG00012
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BG00012 (Experimental): BG00012 administered orally at 120 mg twice daily (BID) for the first 7 days and 240 mg BID thereafter.
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — dimethyl fumarate administered as per the arm description
  Other Names: Tecfidera; DMF; BG00012

SUMMARY:
The primary objective(s) of the study are to assess the BG00012 (dimethyl fumarate) treatment effect on cognition over 2 year period in RRMS patients. The secondary objectives of this study are to further assess BG00012 treatment effect on cognition, predictors of cognitive impairment, clinical efficacy, and patient reported outcomes (PRO): depression, fatigue, quality of life, and work and social life activity.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a confirmed diagnosis of RRMS according to McDonald criteria (Polman, Reingold et al. 2005).
* Must have a baseline EDSS between 0.0 and 5.0, inclusive.
* Must have experienced at least 1 relapse within the 12 months prior to randomization, with a prior brain MRI demonstrating lesion(s) consistent with MS, or show evidence of gadolinium-enhancing lesion(s) of the brain on an MRI performed within the 6 weeks prior to randomization.

Key Exclusion Criteria:

Candidates will be excluded from study entry if any of the following exclusion criteria exist at the time of screening:

* Primary progressive, secondary progressive, or progressive relapsing MS, as defined by Lublin and Reingold (Lublin and Reingold 1996)
* Severe depression (MADRS score >34) (Montgomery and Asberg 1979)
* History of malignancy (except basal cell carcinoma that has been completely excised prior to study enrollment)
* An MS relapse that has occurred within the 30 days prior to inclusion AND/OR the participant has not stabilized from a previous relapse prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with worsening in cognitive improvement over 2 years. | Up to 2 years
  As measured by at least 2 standard deviation (SD) below Italian normative data of the Rao's Brief Repeatable Battery of Neuropsychological Tests (BRB) and a 100-item version of the Stroop Test. The Brief Repeatable Battery of Neuropsychological Tests (BRB-N) is a sensitive measure of cognitive impairment in multiple sclerosis (MS) patients. The Stroop Test is a test used to measure a person's sustained attention for word reading and color naming with and without interference.

SECONDARY OUTCOMES:
Change in cognitive impairment index score (CII) over two years | Up to 2 years
  An individual cognitive change index will be measured by calculating changes on the cognitive impairment index (CII) for each participant between year 0 and year 1, and year 0 and year 2. The CII is an individual cognitive change index aimed at providing a more precise assessment of the amount and direction of cognitive changes over time.
Annualized relapse rate at year 1. | Up to one year
Annualized relapse rate at year 2. | Up to 2 years
Time to relapse over 2 years. | 2 years
Proportion of patients with 6-month sustained progression of disability as measured by at least a 1.0 point increase from a baseline EDSS>1.0 or at least a 1.5 point increase from a baseline EDSS=0). | Up to 2 years
  The Kurtzke Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis. The EDSS quantifies disability in eight Functional Systems (FS) and allows neurologists to assign a Functional System Score (FSS) in each of these. Each functional system is scored on a scale of 0 (no disability) to 5 or 6 (more severe disability). EDSS steps 1.0 to 4.5 refer to people with MS who are fully ambulatory. EDSS steps 5.0 to 9.5 are defined by the impairment to ambulation.
Assessment of baseline demographic, disease characteristics and related patient reported outcomes that predict CI at two years. | Up to 2 years
  Demographics may include age and gender, disease characteristics may include year of diagnosis and disability and PRO may include fatigue and depression at the time of initiation of BG00012.
Change from baseline in a self rating version of the Montgomery and Asberg Depression Rating Scale (MADRS) | 2 years
  The MADRS instrument has nine questions, with an overall score ranging from 0 to 27 points
Change from baseline in fatigue as measured by the Modified Fatigue Impact Scale (MFIS) | 2 years
  The MFIS is a modified form of the Fatigue Impact Scale based on items derived from interviews with MS patients concerning how fatigue impacts their lives. This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items
Change from baseline in Quality of life (QOL) as measured by the EQ-5D Health Survey | 2 years
  The EQ-5D is a widely-used survey instrument for measuring economic preferences for health states. It is a self-administered questionnaire consisting of 5 sets of 3 questions pertaining to specific health states (i.e., mobility, self-care, pain, usual activities, anxiety).
Change from baseline in the Environmental Status Scale (ESS) | 2 years
  The Environmental Status Scale (ESS) is used to quickly evaluate a patient for handicap. It was derived from a measure of socio-economic status. It consists of seven parameters: (1) actual work status, (2) financial and economic status, (3) personal residence or home, (4) personal assistance required, (5) transportation, (6) community services, (7) social activity. Each parameter has a single score from minimum 0 to maximum 5. ESS score is the sum of the points for all 7 parameters: minimum score: 0; maximum score: 35. The higher the score the greater the handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (18):
- Italy (18):
  - Research site, Bari
  - Research site, Cagliari
  - Research site, Catania
  - Research site, Cefalù
  - Research site, Chieti
  - Research site, Ferrara
  - Research site, Fidenza
  - Research site, Florence
  - Research site, Gallarate
  - Research site, Genova
  - Research site, L’Aquila
  - Research site, Milan
  - Research site, Napoli
  - Research site, Orbassano
  - Research site, Padua
  - Research site, Palermo
  - Research site, Pavia
  - Research site, Roma